CLINICAL TRIAL: NCT00003088
Title: A Randomized Phase III Trial of Sequential Chemotherapy Using Doxorubicin, Paclitaxel, and Cyclophosphamide or Concurrent Doxorubicin and Cyclophosphamide Followed by Paclitaxel at 14 or 21 Day Intervals in Women With Node Positive Stage II/IIIA Breast Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9741; U10CA031946 (NIH); CALGB-9741; CDR0000065788 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-09-06 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sequential chemotherapy 21 days (Experimental): Patients received doxorubicin 60 mg/m^2 every 3 weeks for four cycles followed by paclitaxel 175 mg/m^2 every 3 weeks for four cycles followed by cyclophosphamide 600 mg/m^2 every 3 weeks for four cycles.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel
- Concurrent chemotherapy 14 days (Experimental): Patients received doxorubicin 60 mg/m^2 plus cyclophosphamide 600 mg/m^2 every 2 weeks for four cycles followed by paclitaxel 175 mg/m^2 every 2 weeks for four cycles with filgrastim days 3 to 10 of each cycle at 5 µg/kg rounded to either 300 or 480 µg total dose.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel
- Sequential chemotherapy 14 days (Experimental): Patients received doxorubicin 60 mg/m2 every 2 weeks for four cycles followed by paclitaxel 175 mg/m2 every 2 weeks for four cycles followed by cyclophosphamide 600 mg/m2 every 2 weeks for four cycles, with filgrastim days 3 to 10 of each cycle (a total of seven doses) at 5 µg/kg, which could be rounded to either 300 or 480 µg total dose.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel
- Concurrent chemotherapy 21 days (Experimental): Patients received doxorubicin 60 mg/m^2 plus cyclophosphamide 600 mg/m^2 every 3 weeks for four cycles followed by paclitaxel 175 mg/m^2 every 3 weeks for four cycles.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel

INTERVENTIONS:
Drug: cyclophosphamide — given IV
Drug: doxorubicin hydrochloride — given IV
Drug: paclitaxel — given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving drugs at different times or combining more than one drug may kill more tumor cells. It is not yet known which chemotherapy regimen is more effective for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy consisting of either doxorubicin, cyclophosphamide, or paclitaxel given at different times with that of combination chemotherapy consisting of doxorubicin plus cyclophosphamide followed by paclitaxel in treating women with stage II or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the sequential chemotherapy with doxorubicin, paclitaxel and cyclophosphamide to combined doxorubicin and cyclophosphamide followed by paclitaxel for disease free and overall survival in women with node positive stage II or IIIA breast cancer. II. Determine whether increasing the dose density of adjuvant chemotherapy will improve disease free and overall survival. III. Compare the toxicity in patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are randomized into one of four arms (sequential chemotherapy every 2 weeks vs every 3 weeks vs concurrent chemotherapy followed by paclitaxel every 2 weeks vs every 3 weeks). All tumor should be removed by either a modified radical mastectomy or a segmental mastectomy plus axillary node dissection. Adjuvant chemotherapy is started within 84 days following the last surgical procedure. Arm I: Patients receive sequential chemotherapy every 3 weeks. Doxorubicin IV is administered once every 3 weeks for 4 doses. Paclitaxel IV is then administered over 3 hours once every 3 weeks for 4 doses. Cyclophosphamide IV is administered once every 3 weeks for 4 doses following paclitaxel. Arm II: Patients receive sequential chemotherapy every 2 weeks. Doxorubicin IV is administered once every 2 weeks for 4 doses. Paclitaxel IV is then administered over 3 hours once every 2 weeks for 4 doses. Cyclophosphamide IV is administered once every 2 weeks for 4 doses following paclitaxel. Filgrastim (G-CSF) is administered by subcutaneous injection on days 3-10 after each dose of doxorubicin, paclitaxel, and cyclophosphamide. Arm III: Patients receive combination chemotherapy every 3 weeks. Combination doxorubicin IV and cyclophosphamide IV is administered once every 3 weeks for 4 doses. Paclitaxel IV is administered over 3 hours once every 3 weeks for 4 doses following combination chemotherapy. Arm IV: Patients receive combination chemotherapy every 2 weeks. Combination doxorubicin IV and cyclophosphamide IV is administered once every 2 weeks for 4 doses. Paclitaxel IV is administered over 3 hours once every 2 weeks for 4 doses following combination chemotherapy. G-CSF is administered by subcutaneous injection on days 3-10 after each dose of doxorubicin/cyclophophamide and after each dose of paclitaxel. After completion of all chemotherapy, patients receive tamoxifen orally for 5 years. Patients undergo radiotherapy 4-6 weeks after the completion of chemotherapy. Patients are followed every 6 months for 5 years, then annually until death.

PROJECTED ACCRUAL: A total of 2,000 patients will be accrued for this study within 22 months.

ELIGIBILITY:
1. Required Tumor Parameters

   1.1 Patients with operable, histologically confirmed adenocarcinoma of the female breast and positive lymph nodes. Node positivity may be determined by either an axillary node dissection or a positive sentinel node finding by immunohistochemistry or histology. This includes any patient with one or more positive lymph nodes whose tumors are T0, T1, 2 or 3 and N1, N2, MO. Patients with metaplastic carcinoma are eligible. Bilateral disease does not exclude patients from entry.

   1.2 Tumors that are locally advanced at diagnosis are not eligible. This is left to investigator judgment. Patients with tumors fixed to the chest wall, peau d'orange skin changes, skin ulcerations, or clinical inflammatory changes (T4 disease) are excluded from this study. Dermal lymphatic involvement noted on pathology without clinical inflammatory changes will not exclude a patient from this study.

   1.3 Patients with any ERP/PgR status are eligible.
2. Prior treatment:

   2.1 <84 days from mastectomy or within 84 days of axillary dissection if the patient's most extensive breast surgery was a breast sparing procedure.

   2.2 Surgical resection margins - All tumor should be removed by either a modified radical mastectomy or a segmental mastectomy. Node dissection: patients may have had either an axillary node dissection or sentinel lymph node biopsy before beginning treatment on protocol.
   * Mastectomy: There should be no evidence of gross or microscopic tumor at the surgical resection margins noted in the final surgery or pathology reports for patients who have had a modified radical mastectomy. Patients with close margins (tumor < 1 mm from margin) are eligible.
   * Segmental mastectomy (lumpectomy): Although clear margins are preferable, DCIS or LCIS at the surgical resection margin will not render a patient who has undergone a segmental mastectomy ineligible for this study. Invasive tumor at the final resection margin will render a patient ineligible.

   2.3 No prior chemotherapy.

   2.4 No prior radiation therapy for this malignancy. Patients who received radiation to the breast for DCIS are eligible. Patients who have had segmental mastectomy will be treated with radiotherapy according to standard procedures in the treating physician's institution after completion of all chemotherapy. Patients who have had modified radical mastectomy may also receive radiotherapy at the discretion of the treating physician according to institutional guidelines.

   2.5 Patients may receive up to four weeks of tamoxifen therapy for this malignancy and still be eligible for study entry. Patients who received tamoxifen for purposes of chemoprevention (e.g., Breast Cancer Prevention Trial) or for other indications (including previous breast cancer) are eligible. Tamoxifen therapy should be discontinued before the patient is enrolled on this study.
3. Age > 18. There is no upper age limit for enrollment on this study.
4. Required initial laboratory data:

   * Granulocyte count > 1000/mm3
   * Platelet count > 100,000/mm3
   * Bilirubin within upper limits of normal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2005 (Actual)
Dates: Start 1997-09; Primary Completion 2003-04 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc L. Citron, MD, Study Chair — ProHEALTH Care Associates, LLP
Locations (19):
- United States (18):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada

REFERENCES:
- [Background] Muss HB, Berry DA, Cirrincione C, Budman DR, Henderson IC, Citron ML, Norton L, Winer EP, Hudis CA; Cancer and Leukemia Group B Experience. Toxicity of older and younger patients treated with adjuvant chemotherapy for node-positive breast cancer: the Cancer and Leukemia Group B Experience. J Clin Oncol. 2007 Aug 20;25(24):3699-704. doi: 10.1200/JCO.2007.10.9710. PMID 17704418
- [Background] Berry DA, Cirrincione C, Henderson IC, Citron ML, Budman DR, Goldstein LJ, Martino S, Perez EA, Muss HB, Norton L, Hudis C, Winer EP. Estrogen-receptor status and outcomes of modern chemotherapy for patients with node-positive breast cancer. JAMA. 2006 Apr 12;295(14):1658-67. doi: 10.1001/jama.295.14.1658. PMID 16609087
- [Background] Muss H, Berry D, Cirrincione C, et al.: Toxicity of older and younger patients (pts) treated (Rx) with intensive adjuvant chemotherapy (Cx) for node-positive (N+) breast cancer (BC): the CALGB experience. [Abstract] J Clin Oncol 24 (Suppl 18): A-559, 2006.
- [Background] Campone M, Fumoleau P, Bourbouloux E, Kerbrat P, Roche H. Taxanes in adjuvant breast cancer setting: which standard in Europe? Crit Rev Oncol Hematol. 2005 Sep;55(3):167-75. doi: 10.1016/j.critrevonc.2005.04.003. PMID 16039867
- [Background] Orzano JA, Swain SM. Concepts and clinical trials of dose-dense chemotherapy for breast cancer. Clin Breast Cancer. 2005 Dec;6(5):402-11. doi: 10.3816/CBC.2005.n.044. PMID 16381623
- [Background] Berry DA, Cirrincione C, Henderson IC, et al.: Effects of improvements in chemotherapy on disease-free and overall survival of estrogen-receptor negative, node-positive breast cancer: 20-year experience of the CALGB U.S. Breast Intergroup. [Abstract] Breast Cancer Res Treat 88 (Suppl 1): A-29, 2004.
- [Result] Citron ML, Berry DA, Cirrincione C, et al.: Dose-dense (DD) AC followed by paclitaxel is associated with moderate, frequent anemia compared to sequential (S) and/or less DD treatment: update by CALGB on Breast Cancer Intergroup Trial C9741 with ECOG, SWOG, & NCCTG. [Abstract] J Clin Oncol 23 (Suppl 16): A-620, 33s, 2005.
- [Result] Fornier M, Norton L. Dose-dense adjuvant chemotherapy for primary breast cancer. Breast Cancer Res. 2005;7(2):64-9. doi: 10.1186/bcr1007. Epub 2005 Feb 10. PMID 15743513
- [Result] Hudis C, Citron M, Berry D, et al.: Five year follow-up of INT C9741: dose-dense (DD) chemotherapy (CRx) is safe and effective. [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-41, 2005.
- [Result] Schwartz J, Domchek SM, Hwang WT, Fox K. Evaluation of anemia, neutropenia and skin toxicities in standard or dose-dense doxorubicin/cyclophosphamide (AC)-paclitaxel or docetaxel adjuvant chemotherapy in breast cancer. Ann Oncol. 2005 Feb;16(2):247-52. doi: 10.1093/annonc/mdi058. PMID 15668278
- [Result] Citron ML, Berry DA, Cirrincione C, Hudis C, Winer EP, Gradishar WJ, Davidson NE, Martino S, Livingston R, Ingle JN, Perez EA, Carpenter J, Hurd D, Holland JF, Smith BL, Sartor CI, Leung EH, Abrams J, Schilsky RL, Muss HB, Norton L. Randomized trial of dose-dense versus conventionally scheduled and sequential versus concurrent combination chemotherapy as postoperative adjuvant treatment of node-positive primary breast cancer: first report of Intergroup Trial C9741/Cancer and Leukemia Group B Trial 9741. J Clin Oncol. 2003 Apr 15;21(8):1431-9. doi: 10.1200/JCO.2003.09.081. Epub 2003 Feb 13. PMID 12668651
- [Result] Citron M, Berry D, Cirrincione C, et al.: Superiority of dose-dense (DD) over conventional scheduling (CS) and equivalence of sequential (SC) vs. combination adjuvant chemotherapy (CC) for node-positive breast cancer (CALGB 9741, INT C9741). [Abstract] Breast Cancer Res Treat 76 (Suppl 1): A-15, 2002.
- [Derived] Metzger Filho O, Ballman K, Campbell J, Liu M, Ligibel J, Watson M, Chen E, Du L, Stover D, Carey L, Partridge A, Kirshner J, Muss H, Hudis C, Winer EP, Norton L, Symmans WF. Adjuvant Dose-Dense Chemotherapy in Hormone Receptor-Positive Breast Cancer. J Clin Oncol. 2025 Apr;43(10):1229-1239. doi: 10.1200/JCO-24-01875. Epub 2025 Jan 2. PMID 39746162
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/